CLINICAL TRIAL: NCT00234143
Title: A Randomised Controlled Trial of Prolonged Treatment With Darbepoetin Alpha With or Without Recombinant Human Granulocyte Colony Stimulating Factor (G-CSF) Versus Best Supportive Care in Patients With Low-Risk Myelodysplastic Syndromes
Brief Title: Erythropoietin (EPO) and Granulocyte-Colony Stimulating Factor (G-CSF) for Low-Risk Myelodysplastic Syndromes (MDS)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Bartholomew's Hospital (Other)
Responsible Party: Dr. S. Agrawal, St Bartholomew's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04/Q1907/94
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS; EPO; G-CSF; REGiM
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Darbepoetin alfa; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aranesp and Neupogen (Active Comparator): solution for subcutaneous injection , syringe 500 mcg and 300 mcg respectively
  Interventions: Behavioral: Darbepoetin and Filgrastim
- Aranesp (Active Comparator): solution for subcutaneous injection, 500 mcg
  Interventions: Drug: Darbepoetin
- Best supportive care (No Intervention): Red cell transfusion support

INTERVENTIONS:
Behavioral: Darbepoetin and Filgrastim — Aranesp and Neupogen G-CSF (Neupogen) 300 mcg s.c. twice a week, 3-4 days apart and EPO (Aranesp) 500 mcg s.c. once every 2 weeks until week 24, titrate depending of response
  Arms: Aranesp and Neupogen
Drug: Darbepoetin — Aranesp EPO (Aranesp) 500 mcg s.c. once every 2 weeks until 24 weeks, titrate depending of response
  Arms: Aranesp

SUMMARY:
Myelodysplastic syndromes (MDS) are acquired clonal disorders of the bone marrow. The clinical consequences of MDS are bone marrow failure and a predisposition to develop acute myeloid leukaemia (AML). Patients with 'low risk MDS' have less than 10% myeloblasts in the marrow and include the World Health Organization (WHO) subtypes refractory anaemia (RA), refractory anaemia with ring sideroblasts (RARS) and refractory anaemia with excess blasts-I (RAEB-I). This group of patients has a relatively low risk of leukaemic transformation and the major clinical problem is the manifestation of bone marrow failure. Up to 80% of these patients become red cell transfusion dependent. To date, the only curative therapy is allogeneic stem cell transplantation. Unfortunately, a median age at diagnosis of > 65 years excludes this type of therapy for most patients with MDS. The aim of treatment is, therefore, supportive therapy. Long term red cell transfusion therapy carries the problems of acute transfusion reactions: iron overload, alloantibody formation, poor venous access and the risk of transfusion transmitted infection. With time, such patients require increasing frequency of transfusion and obtain decreased length of benefit from transfusion. The quality of life of such patients is significantly reduced. Alternative therapies, therefore, aimed at promoting more effective haemopoiesis and reducing the need for red cell transfusion may improve quality of life, reduce the use of expensive resources such as red cells and iron chelation, and perhaps enhance survival.

Combined darbepoetin alfa (Aranesp) plus G-CSF (Neupogen; filgrastim) in low risk MDS is better than best supportive care, with respect to haemoglobin and quality of life. The study will assess:

* the costs of this approach
* long-term outcomes
* clinical/laboratory parameters allowing early cessation of therapy in patients destined not to respond

DETAILED DESCRIPTION:
STUDY OBJECTIVES:

Primary objectives:

* To compare the Quality of Life of Low-risk MDS patients randomised to receive prolonged treatment with EPO alone, EPO with G-CSF or best supportive care alone.

Secondary objectives:

* To compare the haemoglobin response and transfusion requirements of patients in each of these arms.
* To compare the economics costs of treating patients in each arm, in order to derive a cost:benefit analysis.
* To assess the utility of prognostic factor and predictive factor assessment, in particular against the predictive model proposed by Hellstrom-Lindberg.

STUDY DESIGN:

This trial is a multi-centre, randomised, triple arm, open-label trial of EPO alone (with best supportive care), EPO plus G-CSF (with best supportive care) and best supportive care only in patients with low-risk myelodysplastic syndrome with symptomatic anaemia and/or red cell transfusion dependence. Screening procedures will take place within 42 days of randomisation.

Patients will be randomised in a 1:1:1 ratio to EPO and best supportive care, EPO with G-CSF and best supportive care, or best supportive care only. Patients randomised to drug therapy arms will receive EPO subcutaneously every fortnight ± G-CSF at least weekly, together with red cell transfusions and other supportive care if required. Patients randomised to "best supportive care" only will receive red cell transfusions and supportive care as required. Study visits and selected study investigations will occur every 4 weeks for the first 24 weeks, then at 36 and 52 weeks.

Quality of life (FACT-An and EQ-5D) measures will be used for all arms of the study.

Analysis & Reporting:

Data will be analysed and reported for all endpoints after the final patient has completed the 52 week follow-up.

Data Monitoring Committee:

An independent Data Monitoring Committee (DMC) will ensure the safety of patients enrolled in the trial. This group will be the MRC Leukaemia LDMEC (Chair: Prof. Gordon Murray). The DMC will meet at the commencement of recruitment and will formulate its guidelines for safety and efficacy monitoring. The DMC will provide a report of their meetings to the TSC. The DMC will meet at least annually and more frequently if needed.

Central Morphology Review:

Bone marrow biopsies/aspirates for all patients will be sent for central morphology review to determine eligibility for the study. All screening aspirates and biopsies will be reviewed centrally to confirm the diagnosis of MDS and the categorisation of the WHO/FAB subtype. On-study and end of study bone marrows will also be reviewed. In addition, centralised testing of specialist investigations will be performed.

STUDY ENDPOINTS:

Primary end point:

* Quality of life at 24 weeks (FACT-An & EQ-5D - the latter for use in health economic analyses)

Secondary end points:

* Quality of life at 12, 36 and 52 weeks (FACT-An & EQ-5D)
* Overall erythroid response (major and minor) at 24 weeks (main analysis point) and also at 12 and 52 weeks, as defined by the International Working Group (IWG) criteria
* Incidence of disease progression (i.e. to RAEB or AML)
* Overall survival
* Economic costs of managing anaemia in each arm of the study.

STUDY DURATION:

Patients will be monitored for all study endpoints up to 52 weeks. Patients responding to EPO ± G-CSF will remain on therapy for 52 weeks. Beyond 52 weeks, patients will be followed up indefinitely in order to assess duration of response, incidence of disease progression and overall survival (through the Office of National Statistics).

TOTAL SAMPLE SIZE:

Three hundred & sixty(360) patients, one hundred & twenty (120) in each arm.

DOSING REGIMEN:

The treatment schedule uses the concept of 'frontloading' to give patients the highest doses of EPO at the start of therapy in order to induce a response as quickly as possible. The long-acting nature of darbepoetin alpha avoids excessive frequency of injections, but allows delivery of high doses of EPO. At week 24, if no response is achieved, the study treatment is deemed to have failed and is stopped and patients will receive 'best supportive care' only.

Darbepoetin (120 patients):

* EPO (Aranesp®) 500 mcg s.c. once every 2 weeks.

  1. If a rapid response is obtained (Hb increase > or = 2 g/dl in any 4 week period), titrate down the dose frequency of EPO.
  2. If major response, titrate EPO to lowest dose frequency that maintains the response.
* At 24 weeks :

  1. If no response, stop EPO and give supportive therapy only.
  2. If minor response, continue EPO 500 mcg once every 2 weeks s.c.
  3. If major response, titrate EPO to lowest dose frequency that maintains the response.

Darbepoetine with Filgrastim (120 patients):

* G-CSF (Neupogen®) 300 mcg s.c. twice a week, 3-4 days apart.
* EPO (Aranesp®) 500 mcg s.c. once every 2 weeks.

  1. If a rapid response is obtained (Hb increase > or = 2 g/dl in any 4 week period), titrate down the dose frequency of EPO.
  2. If major response, titrate EPO and G-CSF to lowest dose frequency that maintains the response.
* At 24 weeks :

  1. If no response, stop EPO and G-CSF and give supportive therapy only.
  2. If minor response, continue EPO 500 mcg every 2 weeks s.c. and G-CSF 300 mcg s.c. twice a week, 3-4 days apart.
  3. If major response, titrate EPO and G-CSF to lowest dose frequency that maintains the response.

Best Supportive Care (120 patients):

Patients randomised to no growth factor treatment will receive best supportive care, defined as:

* Red cell transfusion support to achieve a predicted post-transfusion haemoglobin of 11.0 to 12.0 g/dl at a quantity & frequency such that the trough haemoglobin is never < 8.0 g/dl OR

  * such that the patient is never excessively symptomatic, according to local transfusion guidelines/policy.

STUDY DRUG SUPPLIES:

Darbepoetin (Aranesp®) pre-filled syringes 500 mcg and filgrastim (Neupogen®) pre-filled syringes 300 mcg will be supplied by Amgen (UK)and provided free of charge.

SAFETY ASSESSMENTS:

* Vital signs
* Physical examination
* Clinical laboratory assessments
* Concomitant medications
* Adverse events

EFFICACY ASSESSMENTS:

* Quality of life assessments
* Number and frequency of red cell transfusions
* Clinical laboratory assessments
* Bone marrow aspirate assessments

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of MDS - WHO type:

  * refractory anaemia (RA)
  * hypoplastic RA ineligible for or failed immunosuppressive therapy (ALG, cyclosporine)
  * refractory anaemia with ring sideroblasts (RARS)
  * refractory cytopenia with multilineage dysplasia
  * myelodysplastic syndrome unclassifiable
* IPSS low or Int-1, but with BM blasts <5%
* A haemoglobin concentration of < 10g/dl and/or red cell transfusion dependence
* Written informed consent.

Exclusion Criteria:

* MDS with bone marrow blasts ≥5%
* Myelodysplastic syndrome associated with del(5q)(q31-33) syndrome
* Chronic myelomonocytic leukaemia (monocytes >1.0x109/l)
* therapy-related MDS
* Splenomegaly, with spleen ≥ 5 cm from left costal margin
* Platelets <30x109/l
* Uncorrected haematinic deficiency
* Age less than 18 years
* Woman who are pregnant or lactating
* Women of child bearing age unless using reliable contraception
* Life expectancy < 6 months
* Uncontrolled hypertension, previous venous thromboembolism, or uncontrolled cardiac or pulmonary disease
* Previous adverse events to the study medications or its components
* Patients who have had previous therapy with EPO ± G-CSF within 4 weeks of study entry
* Patients currently receiving experimental therapy, e.g. with thalidomide, or who are participating in another clinical trial
* Medical or psychiatric illness, which makes the patient unsuitable or unable to give, informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2004-10

PRIMARY OUTCOMES:
Quality of life (Functional Assessment of Cancer Therapy-Anemia [FACT-An] and EuroQOL-5D [EQ-5D]) | at week 0, 12, 24, 36 and 52

SECONDARY OUTCOMES:
Overall erythroid response (major and minor) at 6 months as defined by the Cheson criteria | week 24
Overall erythroid response (major and minor) at 2 and 12 months as defined by the Cheson criteria | week 8 and 52
Incidence of disease progression (i.e. to RAEB or AML) and overall survival | every 4 weeks until week 24 and at week 36 and 52
Multivariate analysis of prospective laboratory variables in order to generate a prognostic model | every 4 weeks until week 24 and at week 36 and 52
Economic costs of managing anaemia in both arms of the study | every 4 weeks until week 24 and at week 36 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Samir G Agrawal, MD, PhD, Principal Investigator — St. Bartholomew's Hospital
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom